CLINICAL TRIAL: NCT02821910
Title: Relative Bioavailability of Two FDC Tablet Strengths of Empagliflozin/Linagliptin/Metformin Extended Release Compared to the Free Combination of Empagliflozin, Linagliptin and Metformin Extended Release Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: Relative Bioavailability of 2 Fixed Dose Combinations of Empagliflozin/Linagliptin/Metformin Extended Release Compared With Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1361.1; 2015-005082-23 (EudraCT Number)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (3):
- High dose, fed (Experimental): 1 fixed dose combination (FDC) tablet vs. 4 single tablets under fed conditions
  Interventions: Drug: High dose FDC Empagliflozin/Linagliptin/Metformin XR, fed; Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR
- High dose, fasted (Experimental): 1 fixed dose combination (FDC) tablet vs. 4 single tablets under fasted conditions
  Interventions: Drug: High dose FDC Empagliflozin/Linagliptin/Metformin XR, fasted; Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR
- Low dose, fed (Experimental): 1 fixed dose combination (FDC) tablet vs. 4 single tablets under fed conditions
  Interventions: Drug: Low dose FDC Empagliflozin/Linagliptin/Metformin XR, fed; Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR

INTERVENTIONS:
Drug: High dose FDC Empagliflozin/Linagliptin/Metformin XR, fed — High dose Empagliflozin/Linagliptin/Metformin extended release (XR) fixed dose combination (FDC) tablet
  Arms: High dose, fed
Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR — 1x Empagliflozin + 1x Linagliptin + 2x Metformin extended release (XR) tablets
  Arms: High dose, fed
Drug: High dose FDC Empagliflozin/Linagliptin/Metformin XR, fasted — High dose Empagliflozin/Linagliptin/Metformin extended release (XR) fixed dose combination (FDC) tablet
  Arms: High dose, fasted
Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR — 1x Empagliflozin + 1x Linagliptin + 2x Metformin extended release (XR) tablets
  Arms: High dose, fasted
Drug: Low dose FDC Empagliflozin/Linagliptin/Metformin XR, fed — Low dose Empagliflozin/Linagliptin/Metformin extended release (XR) fixed dose combination (FDC) tablet
  Arms: Low dose, fed
Drug: 1 tab Empagliflozin +1 tab Linagliptin +2 tabs Metformin XR — 1x Empagliflozin + 1x Linagliptin + 2x Metformin extended release (XR) tablets
  Arms: Low dose, fed

SUMMARY:
The purpose of this trial is to demonstrate the relative bioavailability of 2 newly developed fixed dose combinations (FDC) tablets containing empagliflozin, linagliptin & metformin extended release (XR) and the single tablets of empagliflozin, linagliptin and metformin XR administered simultaneously.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device Sexually abstinent A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment) Surgically sterilised (including hysterectomy) Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle-stimulating hormone above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including blood pressure, pulse rate or electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The subjects were randomly allocated to the 2 treatment sequences (test (T) - reference (R) or R-T) in 3 separate trial parts. There was a wash-out period of at least 35 days between the treatments.Treatments were administered as single doses in the fed state in Parts 1 and 3, and in the fasted state in Part 2.
Groups:
- FDC 25 Fed (T1)/ E25+L5+M1000 Fed (R1) (Part 1): Subjects were orally administered single dose of 25 milligram (mg) empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 millilitre (mL) of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast
- E25+L5+M1000 Fed (R1)/ FDC 25 Fed (T1) (Part 1): Subjects were orally administered free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered single dose of 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast
- FDC 25 Fast (T2)/ E25+L5+M1000 Fast (R2) (Part 2): Subjects were orally administered single dose of 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after an overnight fast of at least 10 h followed by a wash-out period of at least 35 days and then orally administered free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after an overnight fast of at least 10 h
- E25+L5+M1000 Fast (R2)/ FDC 25 Fast (T2) (Part 2): Subjects were orally administered single dose of free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after an overnight fast of at least 10 h followed by a wash-out period of at least 35 days and then orally administered 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after an overnight fast of at least 10 h
- FDC 10 Fed (T3)/ E10+L5+M1000 Fed (R3) (Part 3): Subjects were orally administered single dose of 10 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered free combination of 10 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast
- E10+L5+M1000 Fed (R3)/ FDC 10 Fed (T3) (Part 3): Subjects were orally administered free combination of 10 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered single dose of 10 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast
Period: Overall Study
Arm/Group | FDC 25 Fed (T1)/ E25+L5+M1000 Fed (R1) (Part 1) | E25+L5+M1000 Fed (R1)/ FDC 25 Fed (T1) (Part 1) | FDC 25 Fast (T2)/ E25+L5+M1000 Fast (R2) (Part 2) | E25+L5+M1000 Fast (R2)/ FDC 25 Fast (T2) (Part 2) | FDC 10 Fed (T3)/ E10+L5+M1000 Fed (R3) (Part 3) | E10+L5+M1000 Fed (R3)/ FDC 10 Fed (T3) (Part 3)
Started | 7 | 8 | 10 | 10 | 7 | 8
Completed | 6 | 8 | 8 | 10 | 7 | 7
Not Completed | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Other than specified | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all randomised subjects, whether treated or not, who were documented to have received at least 1 dose of study drug. This is the full analysis set population in the sense of ICH E9.
Groups:
- Total: Total of all reporting groups
Arm/Group | FDC 25 Fed (T1)/ E25+L5+M1000 Fed (R1) (Part 1) | E25+L5+M1000 Fed (R1)/ FDC 25 Fed (T1) (Part 1) | FDC 25 Fast (T2)/ E25+L5+M1000 Fast (R2) (Part 2) | E25+L5+M1000 Fast (R2)/ FDC 25 Fast (T2) (Part 2) | FDC 10 Fed (T3)/ E10+L5+M1000 Fed (R3) (Part 3) | E10+L5+M1000 Fed (R3)/ FDC 10 Fed (T3) (Part 3) | Total
Number analyzed (Participants) | 7 | 8 | 10 | 10 | 7 | 8 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.9) | 37.1 (11.9) | 36.2 (12.3) | 34.1 (10.0) | 37.3 (11.9) | 35.3 (9.4) | 36.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7 | 2 | 4 | 1 | 21
  Male | 4 | 4 | 3 | 8 | 3 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Empagliflozin in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Concentration (AUC0-tz)
Description: Area under the concentration-time curve of Empagliflozin in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz) is presented.
  Plasma concentrations and/or parameters of a subject were considered as non-evaluable, if for example
  * The subject experienced emesis that occurred at or before 2 times median tmax of the respective treatment (median tmax was to be determined excluding the subject's experiencing emesis)
  * A pre-dose concentration was >5% of the Cmax value measured in that subject
  * Missing samples or concentration data at important phases of PK disposition curve
Time Frame: 1.5 hours (h) before drug administration and 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h,10h, 12h, 24h, 34h, 48h, and 72h after drug administration
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This subject set included all subjects in the TS who provided at least 1 primary or secondary PK parameter that was not excluded according to the criterion's for non-evaluable above.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles (nmol)*hours (h)/litres (L)
Groups:
- FDC 25 Fed (T1): Subjects were orally administered single dose of 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast
- E25+L5+M1000 Fed (R1): Subjects were orally administered single dose of free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast
- FDC 25 Fast (T2): Subjects were orally administered single dose of 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after an overnight fast of at least 10 h
- E25+L5+M1000 Fast (R2): Subjects were orally administered single dose of free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after after an overnight fast of at least 10 h
- FDC 10 Fed (T3): Subjects were orally administered single dose of 10 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast
- E10+L5+M1000 Fed (R3): Subjects were orally administered single dose of free combination of 10 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nanomoles (nmol)*hours (h)/litres (L) | 5990 (25.6) | 6120 (22.8) | 6430 (20.2) | 6250 (18.7) | 2080 (15.4) | 2130 (15.5)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); The statistical model used was an Analysis of variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period', and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; ratio (%) = 96.70, 90% CI 2-sided [92.89 to 100.66], Standard Deviation 5.9 — Relative bioavailability was estimated by the adjusted gMean ratio of T1 divided by R1. Standard deviation is actually intra-individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 100.80, 90% CI 2-sided [97.99 to 103.70], Standard Deviation 4.8 — Relative bioavailability was estimated by the adjusted gMean ratio of T2 divided by R2. Standard deviation is actually intra-individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 99.83, 90% CI 2-sided [95.96 to 103.85], Standard Deviation 5.9 — Relative bioavailability was estimated by the adjusted gMean ratio of T3 divided by R3. Standard deviation is actually intra-individual geometric coefficient variation (gCV)

2. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Concentration (AUC0-tz)
Description: Area under the concentration-time curve of Metformin in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)*h/ milliliter (mL)
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nanograms (ng)*h/ milliliter (mL) | 13900 (29.6) | 13900 (30.9) | 7920 (31.3) | 8260 (33.4) | 12000 (26.0) | 12200 (25.9)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 96.82, 90% CI 2-sided [90.65 to 103.42], Standard Deviation 9.7 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 95.67, 90% CI 2-sided [87.44 to 104.68], Standard Deviation 15.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 98.47, 90% CI 2-sided [92.12 to 105.25], Standard Deviation 9.9 — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Maximum Measured Concentration of Empagliflozin in Plasma (Cmax)
Description: Maximum measured concentration of Empagliflozin in plasma (Cmax) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nmol/L | 594 (17.7) | 630 (20.4) | 872 (24.5) | 817 (31.5) | 232 (20.5) | 235 (18.8)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 94.94, 90% CI 2-sided [86.60 to 104.08], Standard Deviation 13.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 106.63, 90% CI 2-sided [100.65 to 112.96], Standard Deviation 9.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 100.41, 90% CI 2-sided [94.54 to 106.64], Standard Deviation 8.9 — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Maximum Measured Concentration of Metformin in Plasma (Cmax)
Description: Maximum measured concentration of Metformin in plasma (Cmax) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
ng/mL | 1290 (25.0) | 1300 (21.4) | 1010 (31.1) | 1020 (32.8) | 1170 (33.3) | 1150 (32.6)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 97.97, 90% CI 2-sided [91.46 to 104.94], Standard Deviation 10.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 100.04, 90% CI 2-sided [90.23 to 110.91], Standard Deviation 17.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 101.24, 90% CI 2-sided [94.58 to 108.38], Standard Deviation 10.1 — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: Maximum Measured Concentration of Linagliptin in Plasma (Cmax)
Description: Maximum measured concentration of Linagliptin in plasma (Cmax) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nmol/L | 6.37 (20.6) | 6.51 (19.4) | 9.66 (44.5) | 8.35 (27.2) | 6.25 (23.1) | 6.15 (22.8)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 97.50, 90% CI 2-sided [89.94 to 105.71], Standard Deviation 12.0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 117.31, 90% CI 2-sided [103.41 to 133.07], Standard Deviation 22.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 102.74, 90% CI 2-sided [98.56 to 107.10], Standard Deviation 6.2 — [estimate comment as in outcome 1, analysis 3]

6. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72)
Description: Area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 to 72 hours (AUC0-72) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nmol*h/L | 273 (18.7) | 282 (17.2) | 290 (24.7) | 276 (21.1) | 258 (25.1) | 260 (20.2)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 96.34, 90% CI 2-sided [92.13 to 100.75], Standard Deviation 6.6 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 105.07, 90% CI 2-sided [99.95 to 110.45], Standard Deviation 8.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 100.31, 90% CI 2-sided [96.41 to 104.38], Standard Deviation 5.9 — [estimate comment as in outcome 1, analysis 3]

7. Secondary Outcome: Area Under the Concentration-time Curve of the Empagliflozin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the Empagliflozin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nmol*h/L | 6060 (25.7) | 6190 (22.5) | 6490 (20.0) | 6300 (18.7) | 2130 (15.5) | 2180 (15.4)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 96.63, 90% CI 2-sided [92.86 to 100.54], Standard Deviation 5.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 100.87, 90% CI 2-sided [97.96 to 103.86], Standard Deviation 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 99.75, 90% CI 2-sided [95.81 to 103.86], Standard Deviation 6.0 — [estimate comment as in outcome 1, analysis 3]

8. Secondary Outcome: Area Under the Concentration-time Curve of the Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the Metformin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
ng*h/mL | 14100 (29.3) | 14100 (30.0) | 8260 (29.2) | 8600 (33.2) | 12200 (25.8) | 12400 (25.0)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 96.57, 90% CI 2-sided [90.94 to 102.56], Standard Deviation 8.9 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 95.40, 90% CI 2-sided [87.50 to 104.01], Standard Deviation 14.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 98.45, 90% CI 2-sided [92.44 to 104.85], Standard Deviation 9.4 — [estimate comment as in outcome 1, analysis 3]

9. Secondary Outcome: Area Under the Concentration-time Curve of the Linagliptin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the Linagliptin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Number analyzed (Participants) | 15 | 14 | 20 | 18 | 14 | 15
nmol*h/L | 465 (27.2) | 483 (24.8) | 477 (31.1) | 443 (25.2) | 424 (27.6) | 420 (27.1)
Statistical Analysis 1: Comparison: FDC 25 Fed (T1) vs E25+L5+M1000 Fed (R1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 95.08, 90% CI 2-sided [87.36 to 103.48], Standard Deviation 12.6 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FDC 25 Fast (T2) vs E25+L5+M1000 Fast (R2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 105.72, 90% CI 2-sided [98.78 to 113.15], Standard Deviation 11.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: FDC 10 Fed (T3) vs E10+L5+M1000 Fed (R3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio (%) = 101.61, 90% CI 2-sided [92.00 to 112.22], Standard Deviation 14.9 — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: Adverse events occurring up to 168 hours after intake of trial drug administration in each treatment period were assigned to treatment. Adverse events were collected up to 42 days per participant.
Groups:
- E25+L5+M1000 Fast (R2): Subjects were orally administered single dose of free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 tablets of 500 mg metformin extended release tablets with 240 mL of water after after an overnight fast of at least 10 h
- E10+L5+M1000 Fed (R3): Subjects were orally administered single dose of free combination of 10 mg empagliflozin, 5 mg linagliptin and 2 tablets of 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast
Arm/Group | FDC 25 Fed (T1) | E25+L5+M1000 Fed (R1) | FDC 25 Fast (T2) | E25+L5+M1000 Fast (R2) | FDC 10 Fed (T3) | E10+L5+M1000 Fed (R3)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/20 | 0/18 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 4/14 | 6/20 | 4/18 | 1/14 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDC 25 Fed (T1) (N=15) | E25+L5+M1000 Fed (R1) (N=14) | FDC 25 Fast (T2) (N=20) | E25+L5+M1000 Fast (R2) (N=18) | FDC 10 Fed (T3) (N=14) | E10+L5+M1000 Fed (R3) (N=15)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 3 | 3 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blister rupture (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No